CLINICAL TRIAL: NCT00900107
Title: Time Dependent Mobilization of Circulating Progenitor Cells During Strenuous Exercise in Healthy Individuals.
Brief Title: Time-Dependent Mobilization of Circulating Progenitor Cells During Strenuous Exercise in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: University of Jena (Other)
Responsible Party: Principal Investigator, Sven Möbius-Winkler, PD Dr. med., University of Leipzig
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SMW 02
Record Dates: First submitted 2009-05-01; First posted 2009-05-12 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2009-05

CONDITIONS: Healthy Men
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Exercise

SUMMARY:
Only few data are available on the influence of strenuous exercise on the content of circulating progenitor cells and especially the timeframe of their release. The aim of the present study was to investigate the potential influence of 4 hours of cycling on the time-dependent release of progenitor cells.

DETAILED DESCRIPTION:
1. What is the response of hematopoietic and endothelial progenitor cells after a standardized prolonged endurance exercise?
2. What is the kinetic of cell mobilization during this standardized exercise?

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* cardiovascular disease

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Endothelial progenitor cells (EPC) release on | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard C Schuler, Prof. Dr., Study Director — Heart Center Leipzig
Locations (1):
- University Leipzig, Heart Center, Leipzig, Germany